CLINICAL TRIAL: NCT06828198
Title: Open, Non-comparative Study to Evaluate the Effectiveness and Safety of the Medical Device KOS® XL for the Restoration and/or Augmentation of Facial Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Beauty Kozmetik (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGMQUA/0424/MD
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-06

CONDITIONS: Facial Volume
Keywords: restoration and/or augmentation of facial volume

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS® XL (Other): An open, non-comparative, interventional single-armed clinical trial.
  Interventions: Device: KOS® XL

INTERVENTIONS:
Device: KOS® XL — Delivery of medical device as injection

SUMMARY:
The process of facial aging is a result of intricate alterations occurring at both the microscopic and macroscopic levels, leading to changes in facial volume. The observed alterations can be attributed to the process of bone structure resorption, the influence of gravity, redistribution of subcutaneous fat, and injury to the skin. Dermal fillers are utilized for the purpose of enhancing facial features in accordance with the aesthetic ideals of beauty.

KOS® XL in the dermis regulates water balance, osmotic pressure and ion flow and functions as a sieve, excluding certain molecules, enhancing the extracellular domain of cell surfaces and stabilizes skin structures by electrostatic interactions.

The Research Question of the present study is the following: to collect sufficient clinical data to demonstrate compliance with the General Safety and Performance Requirements of KOS® XL when used as intended.

ELIGIBILITY:
Inclusion Criteria:

* Females and males ≥ 22years of age
* Signed informed consent by the subject
* Subject with grade from 3 to 5 on the FVLS.
* Ability to follow study instructions and likely to complete all required visits
* Reliable methods of contraception which result in a low failure rate (i.e. less than 1 % per year) for women of childbearing potential, e.g. implants, injectables, combined oral contraceptives, some intrauterine -devices, sexual abstinence or vasectomized partner) for the entire study duration.

Exclusion Criteria:

1. Using any new over-the-counter or prescription oral or topical, anti-wrinkle products within 30 days before enrolment or planning to begin using such products during the study (Subjects who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study).
2. Subject with a scar, moles or anything on the face which might interfere with the evaluation
3. Subject having received treatment with a laser, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to inclusion
4. Subject having received injection with a resorbable filling product in the face area within the past 18 months prior to inclusion
5. Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …)
6. History of or active autoimmune disease/immune deficiency
7. Suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…)
8. Prone to hypertrophic scars
9. History of allergy to hyaluronic acid or any of the product's components
10. History of allergy to lidocaine or local anaesthesia of amide compounds
11. Known case of porphyria
12. Pregnancy or lactation
13. Taking medications and/or substances known to increase coagulation time (e.g., aspirin, ibuprofen, or herbal supplements) 10 days prior to treatment
14. Have a condition or be in a situation that, in the physician's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
15. Untreated epilepsy
16. Hypersensitivity to gram positive bacterial proteins as hyaluronic acid is produced by Streptococcus type bacteria.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Mean change in facial volume | 6 months
  Mean change in facial volume from baseline on the Facial Volume Loss Scale (FVLS) at month 6 after the last treatment FVLS scale from 1 to 5; where 5 is representing severe indentation of one or more facial regions

SECONDARY OUTCOMES:
Facial Volume Loss Scale (FVLS) | 1, 3 and 12 months
  Change in the FVLS from baseline at 1, 3 and 12 months after the last treatment.
  FVLS scale from 1 to 5; where 5 is representing severe indentation of one or more facial regions
Proportion of participants with at least 1-point improvement on the Facial Volume Loss Scale (FVLS) | 1, 3, 6 and 12 months
  Proportion of participants with at least 1-point improvement from baseline on the FVLS at 1, 3, 6 and 12 months after the last treatment (response rates).
  FVLS scale from 1 to 5; where 5 is representing severe indentation of one or more facial regions
Proportion of participants having a positive aesthetic evolution on the 5-point GAIS | 1, 3, 6 and 12 months
  Proportion of participants having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the physician and subject at 1, 3, 6 and 12 months after the last treatment GAIS scale: from 1 (very much improved) to 5 (worse)
Change from baseline in FACE-Q satisfaction | 1, 3, 6 and 12 months
  Change from baseline in FACE-Q satisfaction with cheekbones and FACE-Q satisfaction with chin at 1, 3, 6 and 12 months after the last treatment FACE-Q satisfaction with cheekbones scale: from 1 (very dissatisfied) to 4 (very satisfied) FACE-Q satisfaction with chin scale: from 1 (very dissatisfied) to 4 (very satisfied)
Short- and long-term adverse effects | 6 and 12 months
  Short- and long-term adverse effects within 2 weeks of the initial or touch-up treatment and during 6, 12 months after the last treatment of the study course, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam D Bayatani, Study Chair
Locations (1):
- Clinica Beyond Dental, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attenello NH, Maas CS. Injectable fillers: review of material and properties. Facial Plast Surg. 2015 Feb;31(1):29-34. doi: 10.1055/s-0035-1544924. Epub 2015 Mar 12. PMID 25763894
- [Background] Mojallal A. Efficacy and Safety of Stylage XL Lidocaine for the Restoration and/or Augmentation of Facial Volume: The Beauty Volume Study. Aesthet Surg J Open Forum. 2023 Jun 26;5:ojad056. doi: 10.1093/asjof/ojad056. eCollection 2023. PMID 37700793